CLINICAL TRIAL: NCT03941535
Title: Comparison of a Decreasing Dose of Daily Intravenous Vitamin K to a Single Dose Given as Standard of Care to an Historical Cohort in Subjects With Larger Burns
Brief Title: Comparison of Vitamin K Doses in Patients With Larger Burn Injuries
Acronym: VITK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joseph M. Still Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMSRF-VITK-P01
Record Dates: First submitted 2019-04-22; First posted 2019-05-08 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Burns
Keywords: Vitamin K
MeSH Terms: conditions — Burns | interventions — Vitamin K

STUDY DESIGN:
Intervention Model Description: Single-center, prospective interventional study to compare a decreasing dose of daily Vitamin K to a matched retrospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decreasing Daily Dose of Vitamin K (Experimental): This group of patients will receive a decreasing dose of Vitamin K IV:
  Days 1-2 = 10mg/day (standard of care) Days 3-4 = 5mg/day Days 5-90 (or date of discharge, death, etc) = 2mg/day
  Interventions: Drug: Vitamin K
- Standard of Care Dose of Vitamin K (Active Comparator): This group of patients will be reviewed retrospectively and would have received Vitamin K IV at 10mg/day during their entire hospital course
  Interventions: Drug: Vitamin K

INTERVENTIONS:
Drug: Vitamin K — Administration of intravenous Vitamin K in doses of 10mg/day, 5mg/day or 2mg/day

SUMMARY:
The use of Vitamin K in treating bleeding diatheses is well documented and accepted as standard of care, as is the effect of Vitamin K on calcium and bone metabolism. In the treatment of larger burns however, there is a paucity of available literature related to optimal daily dosing, goals of therapy and potential complications. This study aims to identify any potential issues arising from the administration of a standard of care dose in an historical cohort of subjects with larger burns to a prospective patient population given a decreasing dose during their intensive care unit (ICU) stay.

DETAILED DESCRIPTION:
This will be a prospective, single-center study. Eligible subjects will present with a minimum 20% Total Body Surface Area (TBSA) burn injury and expected to receive the standard dose of intravenous Vitamin K (10mg/day). Exclusion criteria will include any patient admitted with a history of, or having present at baseline: bleeding disorders, thrombocytopenia, coagulopathy, or liver dysfunction (MELD Score ≥20). Subjects who are moribund, or in the opinion of the investigator, not expected to survive will be excluded, as well as burns induced as a result of a suicide attempt.

The study will enroll approximately 25 subjects in the prospective arm and 25 subjects will be matched from our medical record data base to the basic subject criteria for the chart review portion of the study. Study duration will be 90 days.

The research foundation will request exemption, waiver of HIPAA (Health Insurance Portability and Accountability Act) authorization and waiver of informed consent for the data collection /cohort portion of the study as only burn injury demographics, lab results and dosing regimen will be collected. No protected health information (PHI) will be recorded on patients identified for the cohort arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* The Subject:

  1. is anticipated to be hospitalized for the duration of treatment.
  2. is ≥18 years of age.
  3. or their legally authorized representative is able to provide informed consent.
  4. has been diagnosed with at least 20%TBSA thermal, chemical, or electrical burn.
  5. has a negative urine or serum pregnancy test at screening (if female and has potential for pregnancy)?
  6. is expected to receive the standard of care dosing of intravenous Vitamin K (10g/day).

Exclusion Criteria:

* The Subject:

  1. has a history or, or has present at baseline any of the following:

     1. bleeding disorders
     2. thrombocytopenia
     3. coagulopathy
  2. liver failure (MELD -Model for end stage liver disease score ≥20)
  3. is already therapeutically anticoagulated for PE, DVT, etc.
  4. is participating in another interventional clinical trial for the duration of the study.
  5. is moribund, or in the opinion of the investigator is not expected to survive.
  6. has a burn injury sustained as a result a suicide attempt.

Historical Cohort Inclusion/Exclusion All criteria will be the same except there will be no informed consent requirement. The data collection portion in the historical cohort will be to match burn size, type and etiologies and to collect lab results and other outcomes as specified in the study objectives. No PHI will be collected or shared. Additionally, only patients that received intravenous Vitamin K 10m/day for at least 14 days will be chosen for data collection. Every attempt will be made to match study drug duration (90days) as closely as possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome for the study will be rate of DVT occurrence | 90 days or the study will end at time of discharge or death.
  This outcome will be measured in patients with larger burn % total body surface area (TBSA) burn injury receiving Vitamin K 10mg/day with a decreasing dose over 5 days and maintaining a lower daily dose, versus an historical cohort that received intravenous Vitamin K 10m/day during their entire intensive care unit (ICU) stay.

SECONDARY OUTCOMES:
The secondary outcome for this study will be total number of blood products transfused (Fresh Frozen Plasma - FFP and Packed Red Blood Cells - PRBCs. | 90 days or the study will end at time of discharge or death.
  This outcome will be measured in patients with larger burn % TBSA receiving Vitamin K 10mg/day with a decreasing dose over 5 days and maintaining a lower daily dose, versus an historical cohort that received intravenous Vitamin K 10m/day during their entire ICU stay
The secondary outcome for this study will be comparison of coagulopathy patterns | 90 days or the study will end at time of discharge or death.
  This outcome will be measured in patients with larger burn % TBSA receiving Vitamin K 10mg/day with a decreasing dose over 5 days and maintaining a lower daily dose, versus an historical cohort that received intravenous Vitamin K 10m/day during their entire ICU stay as evidenced by changes in: (Protime - PT, Partial Thromboplastin Time - PTT and International Normalized Ration - INR, liver function abnormalities (Serum glutamic pyruvic transaminase - SGPT, Serum glutamic oxaloacetic transaminase - SGOT, Albumin , Bilirubin).

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events to determine safety and tolerability | from time consent is signed throughout the duration of active study participation (90 days, discharge or death - whichever comes first)
  This outcome will be measured in patients with larger burn % TBSA receiving Vitamin K 10mg/day with a decreasing dose over 5 days and maintaining a lower daily dose, versus an historical cohort that received intravenous Vitamin K 10m/day during their entire ICU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Quinn, MD, Principal Investigator — Joseph M. Still Research Foundation, Inc.
Locations (1):
- Joseph M. Still Burn Center at Doctors Hospital, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zittermann A. Effects of vitamin K on calcium and bone metabolism. Curr Opin Clin Nutr Metab Care. 2001 Nov;4(6):483-7. doi: 10.1097/00075197-200111000-00003. PMID 11706280
- [Background] Fulton RL, McMurdo ME, Hill A, Abboud RJ, Arnold GP, Struthers AD, Khan F, Vermeer C, Knapen MH, Drummen NE, Witham MD. Effect of Vitamin K on Vascular Health and Physical Function in Older People with Vascular Disease--A Randomised Controlled Trial. J Nutr Health Aging. 2016 Mar;20(3):325-33. doi: 10.1007/s12603-015-0619-4. PMID 26892582
- [Background] Yoshida M, Jacques PF, Meigs JB, Saltzman E, Shea MK, Gundberg C, Dawson-Hughes B, Dallal G, Booth SL. Effect of vitamin K supplementation on insulin resistance in older men and women. Diabetes Care. 2008 Nov;31(11):2092-6. doi: 10.2337/dc08-1204. Epub 2008 Aug 12. PMID 18697901
- [Background] Vitamin K Fact Sheet for health professionals. National Institutes of Health Office of Dietary Supplements. U. S. Department of Health and Human Services. Retrieved from https://olds.od.nih.gov/factsheets/VitaminK-HealthProfessional on January 16, 2019.